CLINICAL TRIAL: NCT01304641
Title: Comparison Of Cardiovascular Event Rates In Elderly Patients With Newly Initiated Atorvastatin Or Simvastatin
Brief Title: Cardiovascular Events Based On Statin Initiation In The Elderly
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A2581188
Record Dates: First submitted 2011-02-24; First posted 2011-02-25 (Estimated); Results first posted 2012-04-05 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Cardiovascular; Dyslipidemia
Keywords: Dyslipidemia; Cardiovascular; Statin
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Atorvastatin Initiators
  Interventions: Other: Atorvastatin Initiators
- Simvastatin Initiators
  Interventions: Other: Simvastatin Initiators

INTERVENTIONS:
Other: Atorvastatin Initiators — Retrospective database analysis no intervention performed.
  Groups: Atorvastatin Initiators
Other: Simvastatin Initiators — Retrospective database analysis no intervention performed.
  Groups: Simvastatin Initiators

SUMMARY:
The purpose of this study is to compare rates and risk of primary cardiovascular events among elderly patients newly initiating therapy with atorvastatin or simvastatin. The specific objectives for this project are to: 1) examine the demographic and clinical characteristics of the elderly patients in whom atorvastatin or simvastatin was newly initiated; and 2) compare cardiovascular event rates in elderly patients in whom atorvastatin or simvastatin was newly initiated.

DETAILED DESCRIPTION:
All subjects meeting sample definition, all inclusion criteria, and none of the exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 1 fill for atorvastatin or simvastatin (not including combination therapy) between 01 July 2006 and 30 November 2008
* Age ≥ 65 years as of the year of index date
* Continuous enrollment with medical and pharmacy benefits during the analytic period

Exclusion Criteria:

* 1 or more fills for a statin or other dyslipidemia medication in the 12-month pre-index period
* A pharmacy fill for clopidogrel or nitrates (except concomitant hydralazine) in the 12-month pre-index period
* Patients with evidence of a cardiovascular event in the 12-month pre-index period.
* Patients who received both atorvastatin and simvastatin on the index date
* Patients with unknown gender or region
* Patients who received dyslipidemia medications other than the index drug within 1 months (30 days) following the index date

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: This study included commercial health plan members and Medicare Advantage Part D enrollees ages 65 years and older with a prescription for atorvastatin or simvastatin filled between 01 July 2006 and 30 November 2008 (subject identification period). The first observed atorvastatin or simvastatin fill during the subject identification period was defined as the index drug and the fill date was defined as the index date. A 12-month period prior to the index date (defined as the pre-index period) was used for identification of comorbid exclusionary conditions. The 12-month period prior to index date was also used for assessment of pre-index patient characteristics. Patients were observed for a minimum of 3 months (following index date) until the earlier of either 1) disenrollment from the health plan or 2) 28 February 2009 (post-index period). The pre- and post-index periods in combination were defined as the analytic period.
Sampling Method: Non-Probability Sample
Enrollment: 31603 (Actual)
Dates: Start 2009-11; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2581188&StudyName=Cardiovascular%20Events%20Based%20On%20Statin%20Initiation%20In%20The%20Elderly

RESULTS

PARTICIPANT FLOW:
Groups:
- Atorvastatin: Participants who had been on atorvastatin with dose strength ranging from 10 milligram (mg) to 80 mg were observed for 12 months and a 3 month follow-up period.
- Simvastatin: Participants who had been on simvastatin with dose strength ranging from 5 mg to 80 mg were observed for 12 months and a 3 month follow-up period.
Period: Overall Study
Arm/Group | Atorvastatin | Simvastatin
Started | 11470 | 20132
Completed | 11470 | 20132
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atorvastatin | Simvastatin | Total
Number analyzed (Participants) | 11470 | 20132 | 31602
Age, Customized [Number; unit: Participants]
  65 to 74 years | 8008 | 13369 | 21377
  75 to 84 years | 2937 | 5790 | 8727
  Greater than and equal to (>=) 85 years | 525 | 973 | 1498
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6922 | 12070 | 18992
  Male | 4548 | 8062 | 12610

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Post-index Cardiovascular (CV) Events
Description: CV events were defined as an inpatient or emergency department admission for heart failure (HF), myocardial infarction (MI), ischemic heart disease (IHD), cerebrovascular disease, peripheral vascular disease (PVD), aortic aneurysm, and/or revascularization. CV events were identified using medical claims.
Time Frame: At least 3 months from the post-index date (baseline) or end of study (28 February 2009)
Population: Evaluable analysis population included all participants who met inclusion criteria.
Measure: Number; unit: Participants
Arm/Group | Atorvastatin | Simvastatin
Number analyzed (Participants) | 11470 | 20132
Participants | 700 | 1012
Statistical Analysis 1: Comparison: Atorvastatin vs Simvastatin; Test type: Superiority or Other; p < 0.001, Chi-squared

2. Primary Outcome: Hazard Ratio for First Cardiovascular (CV) Event
Description: Hazard ratio of atorvastatin versus simvastatin for first CV event. Hazard ratio of atorvastatin versus simvastatin was obtained from a Cox proportional hazards model.
Time Frame: At least 3 months from the post-index date (baseline) or end of study (28 February 2009)
Population: Evaluable analysis population included all participants who met inclusion criteria.
Measure: Number; unit: Participants
Arm/Group | Atorvastatin | Simvastatin
Number analyzed (Participants) | 11470 | 20132
Participants
  Number of participants with event | 700 | 1012
  Number of participants without event | 10770 | 19120
Statistical Analysis 1: Comparison: Atorvastatin vs Simvastatin; Test type: Superiority or Other; p = 0.140, Regression, Cox; Hazard Ratio (HR) = 1.078, 95% CI 2-sided [0.976 to 1.192]

3. Secondary Outcome: Low-density Lipoprotein Cholesterol (LDL-C)
Time Frame: At least 3 months from the post-index date (baseline) or end of study (28 February 2009)
Population: Evaluable analysis population included all participants who met inclusion criteria. Here, the 'N' (number of participants analyzed) is signifying those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: milligram/deciliter (mg/dL)
Arm/Group | Atorvastatin | Simvastatin
Number analyzed (Participants) | 887 | 1678
milligram/deciliter (mg/dL) | 94.07 (24.50) | 98.03 (25.56)
Statistical Analysis 1: Comparison: Atorvastatin vs Simvastatin; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

4. Secondary Outcome: Mean Dose
Description: The first observed study medication fill during the participation identification period was defined as the index drug. The initial dose of the index drug was determined based on the pharmacy claims.
Time Frame: At least 3 months from the post-index date (baseline) or end of study (28 February 2009)
Population: Evaluable analysis population included all participants who met inclusion criteria.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Atorvastatin | Simvastatin
Number analyzed (Participants) | 11470 | 20132
mg | 19.46 (15.91) | 28.36 (18.60)
Statistical Analysis 1: Comparison: Atorvastatin vs Simvastatin; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

5. Secondary Outcome: Number of Participants Per Dose
Description: Index dose was categorized as low dose (atorvastatin 10 mg, simvastatin up to 20 mg), medium dose (atorvastatin 20 mg, simvastatin 40 mg), and high dose (atorvastatin 40 or 80 mg, simvastatin 80 mg).
Time Frame: At least 3 months from the post-index date (baseline) or end of study (28 February 2009)
Population: Evaluable analysis population included all participants who met inclusion criteria.
Measure: Number; unit: Participants
Arm/Group | Atorvastatin | Simvastatin
Number analyzed (Participants) | 11470 | 20132
Participants
  Low dose | 5639 | 12344
  Medium dose | 3940 | 6768
  High dose | 1891 | 1020
Statistical Analysis 1: Comparison: Atorvastatin vs Simvastatin; Test type: Superiority or Other; p < 0.001, Chi-squared

6. Secondary Outcome: Length of Post-index Period
Description: Post-index period included time during which participants were observed for a minimum of 3 months following index date (fill date on which first observed atorvastatin or simvastatin was filled during the participant identification period) until disenrollment or end of study treatment (28 February 2009).
Time Frame: Index date (baseline) up to end of study (28 February 2009)
Population: Evaluable analysis population included all participants who met inclusion criteria.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Atorvastatin | Simvastatin
Number analyzed (Participants) | 11470 | 20132
Days | 519.10 (251.38) | 448.41 (238.11)
Statistical Analysis 1: Comparison: Atorvastatin vs Simvastatin; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

7. Secondary Outcome: Percentage of Participants Who Adhered to Index Therapy
Description: Percentage of participants who adhered to index therapy was evaluated. Treatment adherence was defined as the number of days covered by index medication divided by the number of days in the post-index period, expressed as a percentage.
Time Frame: At least 3 months from the post-index date (baseline) or end of study (28 February 2009)
Population: Evaluable analysis population included all participants who met inclusion criteria.
Measure: Number; unit: Percentage of participants
Arm/Group | Atorvastatin | Simvastatin
Number analyzed (Participants) | 11470 | 20132
Percentage of participants
  Less than 80 percent | 64.92 | 57.32
  Greater than or equal to 80 percent | 35.08 | 42.68
Statistical Analysis 1: Comparison: Atorvastatin vs Simvastatin; Test type: Superiority or Other; p < 0.001, Chi-squared

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study. As it was a retrospective study, safety data was not analyzed.
Arm/Group | Atorvastatin | Simvastatin
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.